CLINICAL TRIAL: NCT00775970
Title: Influence of Walking on Spontaneous Physical Activity and on Lipid Oxidation Following Dietary Treatment of Obesity
Brief Title: Walking, Spontaneous Physical Activity and Lipid Oxidation After Dietary Treatment of Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital, Tours, University Hospital, Tours
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PHRI07-DJ APS
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Obesity
Keywords: Obesity; Weight loss maintenance; Spontaneous physical activity; Lipid oxydation; Walking
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: walking activity

SUMMARY:
The purpose of this study is to determine whether walking exercise after dietary treatment of obesity is associated with a decrease of the daily spontaneous physical activity and\or with an increase of the time spent in sedentary activities. Our hypothesis is that the practice of walking as an exercise during the phase of weight stability following the dietary treatment of obesity leads to a reduction of spontaneous physical activity and\or to an increase in the time spent in sedentary activities.

DETAILED DESCRIPTION:
The subjects of this study will be randomised in 2 groups:

A group with usual follow-up and a group with usual follow-up associated with recommendations to introduce a program of walking achieving gradually 2000-2500 kcal/week.

ELIGIBILITY:
Inclusion Criteria:

* Women from 18 to 50 year-old
* In phase of weight stability
* BMI<40kg/m²

Exclusion Criteria:

* History of bariatric surgery
* Diabetes
* Suspicion of obstructive sleep apnea syndrome

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-05

PRIMARY OUTCOMES:
Daily time of moderate physical activity, inactivity and total physical activity measured by a portable monitor of physical activity | 10 weeks

SECONDARY OUTCOMES:
Daily energy expenditure and respiratory quotient during a stay in a respiration chamber | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David JACOBI, MD, Principal Investigator — Service de médecine Interne-Nutrition
Locations (1):
- Service de Médecine Interne - Nutrition / CHRU de Tours, Tours, France

REFERENCES:
- [Background] Brage S, Brage N, Franks PW, Ekelund U, Wong MY, Andersen LB, Froberg K, Wareham NJ. Branched equation modeling of simultaneous accelerometry and heart rate monitoring improves estimate of directly measured physical activity energy expenditure. J Appl Physiol (1985). 2004 Jan;96(1):343-51. doi: 10.1152/japplphysiol.00703.2003. Epub 2003 Sep 12. PMID 12972441
- [Background] Fogelholm M, Kukkonen-Harjula K. Does physical activity prevent weight gain--a systematic review. Obes Rev. 2000 Oct;1(2):95-111. doi: 10.1046/j.1467-789x.2000.00016.x. PMID 12119991
- [Background] Froidevaux F, Schutz Y, Christin L, Jequier E. Energy expenditure in obese women before and during weight loss, after refeeding, and in the weight-relapse period. Am J Clin Nutr. 1993 Jan;57(1):35-42. doi: 10.1093/ajcn/57.1.35. PMID 8416662
- [Background] Jequier E, Schutz Y. Long-term measurements of energy expenditure in humans using a respiration chamber. Am J Clin Nutr. 1983 Dec;38(6):989-98. doi: 10.1093/ajcn/38.6.989. PMID 6650455
- [Background] Kraemer WJ, Volek JS, Clark KL, Gordon SE, Incledon T, Puhl SM, Triplett-McBride NT, McBride JM, Putukian M, Sebastianelli WJ. Physiological adaptations to a weight-loss dietary regimen and exercise programs in women. J Appl Physiol (1985). 1997 Jul;83(1):270-9. doi: 10.1152/jappl.1997.83.1.270. PMID 9216973
- [Background] Levine JA, Eberhardt NL, Jensen MD. Role of nonexercise activity thermogenesis in resistance to fat gain in humans. Science. 1999 Jan 8;283(5399):212-4. doi: 10.1126/science.283.5399.212. PMID 9880251
- [Background] Levine JA, Schleusner SJ, Jensen MD. Energy expenditure of nonexercise activity. Am J Clin Nutr. 2000 Dec;72(6):1451-4. doi: 10.1093/ajcn/72.6.1451. PMID 11101470
- [Background] Nicklas BJ, Rogus EM, Goldberg AP. Exercise blunts declines in lipolysis and fat oxidation after dietary-induced weight loss in obese older women. Am J Physiol. 1997 Jul;273(1 Pt 1):E149-55. doi: 10.1152/ajpendo.1997.273.1.E149. PMID 9252491
- [Background] van Aggel-Leijssen DP, Saris WH, Hul GB, van Baak MA. Short-term effects of weight loss with or without low-intensity exercise training on fat metabolism in obese men. Am J Clin Nutr. 2001 Mar;73(3):523-31. doi: 10.1093/ajcn/73.3.523. PMID 11237927
- [Background] van Aggel-Leijssen DP, Saris WH, Wagenmakers AJ, Hul GB, van Baak MA. The effect of low-intensity exercise training on fat metabolism of obese women. Obes Res. 2001 Feb;9(2):86-96. doi: 10.1038/oby.2001.11. PMID 11316351
- [Background] Zurlo F, Lillioja S, Esposito-Del Puente A, Nyomba BL, Raz I, Saad MF, Swinburn BA, Knowler WC, Bogardus C, Ravussin E. Low ratio of fat to carbohydrate oxidation as predictor of weight gain: study of 24-h RQ. Am J Physiol. 1990 Nov;259(5 Pt 1):E650-7. doi: 10.1152/ajpendo.1990.259.5.E650. PMID 2240203